CLINICAL TRIAL: NCT04136184
Title: A Phase 3 Global, Open-Label, Randomized Study to Evaluate the Efficacy and Safety of ION-682884 in Patients With Hereditary Transthyretin-Mediated Amyloid Polyneuropathy
Brief Title: NEURO-TTRansform: A Study to Evaluate the Efficacy and Safety of Eplontersen (Formerly Known as ION-682884, IONIS-TTR-LRx and AKCEA-TTR-LRx) in Participants With Hereditary Transthyretin-Mediated Amyloid Polyneuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ION-682884-CS3; 2019-001698-10 (EudraCT Number)
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Hereditary Transthyretin-Mediated Amyloid Polyneuropathy
Keywords: Polyneuropathy; Amyloidosis; ATTR; TTR
MeSH Terms: conditions — Polyneuropathies; Amyloidosis | interventions — Inotersen; eplontersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Inotersen (Active Comparator): Participants received inotersen, 300 milligrams (mg), subcutaneously (SC), once weekly up to Week 34. After Week 35 assessment, participants received eplontersen, 45 mg, SC, once every 4 weeks starting from Week 37 up to Week 81.
  Interventions: Drug: Inotersen; Drug: Eplontersen
- Eplontersen (Experimental): Participants received eplontersen, 45 mg, SC, once every 4 weeks up to Week 81.
  Interventions: Drug: Eplontersen

INTERVENTIONS:
Drug: Inotersen — Inotersen by subcutaneous injection
  Other Names: TEGSEDI; ISIS 420915
  Arms: Inotersen
Drug: Eplontersen — Eplontersen by subcutaneous injection
  Other Names: ION-682884; AKCEA-TTR-LRx; IONIS-TTR-LRx

SUMMARY:
The main objective of this study was to evaluate the efficacy of eplontersen as compared with the historical control of the placebo cohort in the NEURO-TTR trial (NCT01737398/2012-001831-30), in subjects with hereditary transthyretin-mediated amyloidosis polyneuropathy (hATTR-PN). For more information, please visit http://www.neuro-ttransform.com/.

DETAILED DESCRIPTION:
This study was a multicenter, open-label study in up to 168 participants, who were randomized to receive subcutaneous (SC) injections of either eplontersen once every 4 weeks or inotersen once a week. Participants also received daily supplemental doses of the recommended daily allowance of vitamin A. Participants included in the inotersen reference arm crossed over to eplontersen at Week 37 after completing the Week 35 assessments.

ELIGIBILITY:
Key Inclusion Criteria:

1. Aged 18 to 82 years at the time of informed consent
2. Females must be non-pregnant and non-lactating, and either surgically sterile or post-menopausal or abstinent
3. Males must be surgically sterile or, abstinent or, if engaged in sexual relations with a woman of child-bearing potential, the participant or the participantss non-pregnant female partner must be using a highly effective contraceptive method
4. Diagnosis of hereditary transthyretin-mediated polyneuropathy as defined by meeting all 3 of the following:

   * Stage 1 or Stage 2 Familial Amyloid Polyneuropathy (FAP) or Coutinho Stage
   * Documented genetic mutation in the TTR gene
   * Symptoms and signs consistent with neuropathy associated with transthyretin amyloidosis, including Neuropathy Impairment Score (NIS) ≥ 10 and ≤ 130

Key Exclusion Criteria:

1. Clinically-significant (CS) abnormalities in medical history, screening laboratory results, physical or physical examination that would render a participants unsuitable for inclusion, including but not limited to abnormal safety labs
2. Karnofsky performance status ≤ 50
3. Other causes of sensorimotor or autonomic neuropathy (e.g., autoimmune disease), including uncontrolled diabetes
4. Prior liver transplant or anticipated liver transplant within 1-yr of Screening
5. New York Heart Association (NYHA) functional classification of ≥ 3
6. Acute coronary syndrome within 6 months of screening or major surgery within 3 months of Screening
7. Other types of amyloidosis
8. Have any other conditions, which, in the opinion of the Investigator or Sponsor would make the participant unsuitable for inclusion, or could interfere with the participant participating in or completing the Study
9. Current treatment with any approved drug for hereditary TTR amyloidosis such as Vyndaqel® / Vyndamax™ (tafamidis), Tegsedi™ (inotersen), Onpattro™ (patisiran), off-label use of diflunisal or doxycycline, and tauroursodeoxycholic acid (TUDCA). If previously treated with Vyndaqel® / Vyndamax™, diflunisal or doxycycline, and TUDCA, must have discontinued treatment for at least 2 weeks prior to Study Day 1
10. Previous treatment with Tegsedi™ (Inotersen) or Onpattro™ (patisiran), or other oligonucleotide or RNA therapeutic (including siRNA)

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (45):
- United States (12):
  - Mayo Clinic - Arizona, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Indiana University School of Medicine - Indianapolis, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University Neurology Research Office, Baltimore, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - The Neurological Institute of New York, New York, New York
  - University of North Carolina Hospitals - Neurology Clinic, Chapel Hill, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - University of Washington Medical Center, Seattle, Washington
- Argentina (4):
  - Hospital Italiano de Buenos Aires, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Hospital El Cruce, San Juan Bautista, Buenos Aires
  - STAT Research, Buenos Aires
  - Instituto Fleni, Buenos Aires
- Perron Institute for Neurological and Translational Science, Nedlands, Western Australia, Australia
- Brazil (5):
  - Instituto de Neurologia de Curitiba, Curitiba, Paraná
  - Universidade Estadual de Campinas, Campinas
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, Ribeirão Preto
  - Hospital Universitário Clementino Fraga Filho, Rio de Janeiro
  - Associação de Assistência à Criança Deficiente - Unidade Lar Escola, São Paulo
- Toronto General Hospital, Toronto, Ontario, Canada
- The Cyprus Institute of Neurology and Genetics, Égkomi, Cyprus
- France (3):
  - Centre Hospitalier Universitaire de Toulouse, Toulouse, Haute-Garonne
  - Hôpital de la Timone, Marseille
  - Hôpital Bicêtre, Le Kremlin-Bicêtre, Île-de-France Region
- Germany (2):
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Universitätsklinikum Heidelberg, Heidelberg
- University General Hospital of Heraklion (PAGNI), Heraklion, Crete, Greece
- Italy (4):
  - Azienda Ospedaliera Universitaria Policlinico Gaetano Martino, Messina
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
- Auckland City Hospital, Grafton, Auckland, New Zealand
- Portugal (2):
  - Centro Hospitalar Universitário Lisboa Norte - Hospital De Santa Maria, Lisbon
  - Centro Hospitalar Universitário do Porto - Hospital Geral de Santo Antonio, Porto
- Spain (2):
  - Hospital Son Llàtzer, Palma de Mallorca, Balearic Islands
  - Hospital Clínico San Carlos, Madrid
- Norrlands Universitetssjukhus, Umeå, Sweden
- Taiwan (4):
  - Chang Gung Memorial Hospital - Linkou Branch, Taoyuan, Guishan District
  - China Medical University Hospital, Taichung, Taichung
  - Taipei Veterans General Hospital, Taipei City, Taipei
  - National Taiwan University Hospital, Taipei
- İstanbul Üniversitesi - Istanbul Tıp Fakültesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Coelho T, Marques W Jr, Dasgupta NR, Chao CC, Parman Y, Franca MC Jr, Guo YC, Wixner J, Ro LS, Calandra CR, Kowacs PA, Berk JL, Obici L, Barroso FA, Weiler M, Conceicao I, Jung SW, Buchele G, Brambatti M, Chen J, Hughes SG, Schneider E, Viney NJ, Masri A, Gertz MR, Ando Y, Gillmore JD, Khella S, Dyck PJB, Waddington Cruz M; NEURO-TTRansform Investigators. Eplontersen for Hereditary Transthyretin Amyloidosis With Polyneuropathy. JAMA. 2023 Oct 17;330(15):1448-1458. doi: 10.1001/jama.2023.18688. PMID 37768671
- [Derived] Coelho T, Waddington Cruz M, Chao CC, Parman Y, Wixner J, Weiler M, Barroso FA, Dasgupta NR, Jung SW, Schneider E, Viney NJ, Dyck PJB, Ando Y, Gillmore JD, Khella S, Gertz MA, Obici L, Berk JL. Characteristics of Patients with Hereditary Transthyretin Amyloidosis-Polyneuropathy (ATTRv-PN) in NEURO-TTRansform, an Open-label Phase 3 Study of Eplontersen. Neurol Ther. 2023 Feb;12(1):267-287. doi: 10.1007/s40120-022-00414-z. Epub 2022 Dec 16. PMID 36525140
- [Derived] Coelho T, Ando Y, Benson MD, Berk JL, Waddington-Cruz M, Dyck PJ, Gillmore JD, Khella SL, Litchy WJ, Obici L, Monteiro C, Tai LJ, Viney NJ, Buchele G, Brambatti M, Jung SW, St L O'Dea L, Tsimikas S, Schneider E, Geary RS, Monia BP, Gertz M. Design and Rationale of the Global Phase 3 NEURO-TTRansform Study of Antisense Oligonucleotide AKCEA-TTR-LRx (ION-682884-CS3) in Hereditary Transthyretin-Mediated Amyloid Polyneuropathy. Neurol Ther. 2021 Jun;10(1):375-389. doi: 10.1007/s40120-021-00235-6. Epub 2021 Feb 26. PMID 33638113

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 46 investigative sites in 15 countries (Argentina, Australia, Brazil, Canada, Cyprus, France, Germany, Italy, New Zealand, Portugal, Spain, Sweden, Taiwan, Turkey, and the United States) from 11 December 2019 to 12 July 2023.
Pre-assignment Details: Participants with a diagnosis of hereditary transthyretin-mediated amyloid Polyneuropathy (hATTR-PN) were randomized in a 6:1 ratio to receive eplontersen (ION-682884) or inotersen respectively. As pre-specified in the protocol, the placebo-cohort group from ISIS 420915-CS2 (NEURO-TTR) study (NCT01737398-3), which was used as an external control for efficacy analysis in this study.
Period: Overall Study
Arm/Group | Inotersen | Eplontersen
Started | 24 | 144
Completed | 1 | 22
Not Completed | 23 | 122
Not completed — Lost to Follow-up | 0 | 3
Not completed — Voluntary Withdrawal (including enrolled OLE) | 23 | 119

BASELINE CHARACTERISTICS:
Population: Randomized set included participants who were screened and who received a randomization assignment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Inotersen | Eplontersen | Total
Number analyzed (Participants) | 24 | 144 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (14.38) | 53.0 (15.00) | 52.8 (14.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 44 | 52
  Male | 16 | 100 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 22 | 27
  Not Hispanic or Latino | 18 | 120 | 138
  Unknown or Not Reported | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 22 | 24
  Black or African American | 0 | 5 | 5
  White | 19 | 112 | 131
  Other | 2 | 3 | 5
  Multiple | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2
Serum Transthyretin (TTR) Concentration [Mean (Standard Deviation); unit: grams per litre (g/L)] | 0.22 (0.069) | 0.23 (0.075) | 0.23 (0.074)
Modified Neuropathy Impairment Score Plus 7 (mNIS+7) Composite Score [Mean (Standard Deviation); unit: scores on a scale] — The mNIS+7 composite score is a measure of neurologic impairment that evaluates muscle weakness, sensation, reflexes, nerve conduction, and autonomic function. The mNIS+7 consists of 2 composite scores: the NIS composite score (maximum of 244 points) and the modified +7 composite score (maximum of 102.32 points). The mNIS+7 composite total score has a range of -22.32 to 346.32, and a higher score indicates lower function.
  scores on a scale | 65.06 (33.515) | 81.28 (43.401) | 78.97 (42.43)
Norfolk Quality of Life Diabetic Neuropathy (QoL-DN) Total Score [Mean (Standard Deviation); unit: scores on a scale] — The Norfolk QoL-DN score is a measure of physical function/large fiber neuropathy, symptoms, activities of daily living, small fiber neuropathy, and autonomic neuropathy. The Norfolk QoL-DN total score has a range of -4 to 138, and a higher score indicates poorer quality of life. Population: Randomized set included participants who were screened and who received a randomization assignment. Number analyzed is the number of participants with data available for analysis.
  scores on a scale
    number analyzed (Participants) | 24 | 137 | 161
    (all) | 40.05 (21.488) | 44.09 (26.590) | 43.49 (25.87)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Modified Neuropathy Impairment Score Plus 7 (mNIS+7) at Week 66
Description: mNIS+7 composite score is a measure of neurologic impairment evaluating muscle weakness, sensation, reflexes, nerve conduction, and autonomic function. mNIS+7 consists of 2 composite scores: the NIS composite score (maximum of 244 points) & the modified +7 composite score (maximum of 102.32 points). mNIS+7 composite total score range= -22.32 to 346.32. Higher score indicated a lower function. Least square (LS) mean & standard error (SE) were analyzed using Mixed Effects Model with Repeated Measures (MMRM). As pre-specified in the protocol, the efficacy of eplontersen was to be assessed by comparing participants enrolled in the eplontersen arm only with the external placebo group. There was no statistical comparison planned between the inotersen arm and the eplontersen-treated/external placebo group arms.
Time Frame: Baseline, Week 66
Population: FAS: all randomized participants who received at least 1 injection of ION-682884/inotersen & had a baseline & 1 post-baseline efficacy assessment for mNIS+7 score/Norfolk QOL-DN questionnaire total score. NEURO-TTR, FAS: all randomized participants who received at least 1 injection of study drug & had a baseline & 1 post-baseline efficacy assessment for the mNIS+7 or Norfolk QOL-DN questionnaire total score. Overall number analyzed = number of participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Groups:
- External Placebo: Participants in the external placebo arm received 3 SC doses of placebo during Week 1, followed by once-weekly SC administration for 64 weeks of the NEURO-TTR study.
Arm/Group | Eplontersen | External Placebo
Number analyzed (Participants) | 128 | 52
scores on a scale | 0.2964 (2.4123) | 25.0557 (2.3874)
Statistical Analysis 1: Comparison: Eplontersen vs External Placebo; Test type: Superiority; p = 0.00000001, MMRM; Difference in LS Mean = -24.7593, 95% CI 2-sided [-30.9552 to -18.5635]

2. Primary Outcome: Change From Baseline in the Norfolk Quality of Life Diabetic Neuropathy (QoL-DN) Questionnaire at Week 66
Description: The Norfolk QoL-DN score is a measure of physical function/large fiber neuropathy, symptoms, activities of daily living, small fiber neuropathy, and autonomic neuropathy. The Norfolk QoL-DN total score has a range of -4 to 138, and a higher score indicates poorer quality of life. LS mean and SE were analyzed using MMRM. As pre-specified in the protocol, the efficacy of eplontersen was to be assessed by comparing participants enrolled in the eplontersen arm only with the external placebo group. There was no statistical comparison planned between the inotersen arm and the eplontersen-treated/external placebo group arms.
Time Frame: Baseline, Week 66
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Eplontersen | External Placebo
Number analyzed (Participants) | 128 | 52
scores on a scale | -5.4964 (2.2976) | 14.2388 (2.3488)
Statistical Analysis 1: Comparison: Eplontersen vs External Placebo; Test type: Superiority; p = 0.00000001, MMRM; Difference in LS Mean = -19.7352, 95% CI 2-sided [-25.6301 to -13.8403]

3. Primary Outcome: Percent Change From Baseline in Serum TTR Concentration at Week 65
Description: As pre-specified in the protocol, the efficacy of eplontersen was to be assessed by comparing participants enrolled in the eplontersen arm only with the external placebo group. There was no statistical comparison planned between the inotersen arm and the eplontersen-treated/external placebo group arms. Overall number analyzed is the number of participants with data available for analysis.
Time Frame: Baseline, Week 65
Population: FAS was defined as all randomized participants who received at least 1 injection of ION-682884/inotersen and had a baseline & at least 1 post-baseline efficacy assessment for mNIS+7 score or Norfolk QOL-DN questionnaire total score. For NEURO-TTR trial, FAS included all randomized participants who received at least 1 injection of study drug and had a baseline and at least 1 post-baseline efficacy assessment for the mNIS+7 score or Norfolk QOL-DN questionnaire total score.
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Eplontersen | External Placebo
Number analyzed (Participants) | 135 | 51
percentage | -81.65 (1.605) | -11.24 (1.910)
Statistical Analysis 1: Comparison: Eplontersen vs External Placebo; Test type: Superiority; p = 0.00000001, MMRM; Difference in LS Mean = -70.42, 95% CI 2-sided [-75.17 to -65.66]

4. Primary Outcome: Percent Change From Baseline in Serum TTR Concentration at Week 35
Description: as for outcome 3
Time Frame: Baseline, Week 35
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Eplontersen | External Placebo
Number analyzed (Participants) | 139 | 57
percentage | -81.14 (1.674) | -14.49 (1.966)
Statistical Analysis 1: Comparison: Eplontersen vs External Placebo; Test type: Superiority; p = 0.00000001, MMRM; Difference in LS Mean = -66.65, 95% CI 2-sided [-71.59 to -61.71]

5. Primary Outcome: Change From Baseline in Modified Neuropathy Impairment Score Plus 7 (mNIS+7) at Week 35
Description: mNIS+7 composite score is a measure of neurologic impairment evaluating muscle weakness, sensation, reflexes, nerve conduction, and autonomic function. mNIS+7 consists of 2 composite scores: NIS composite score (maximum of 244 points) & the modified +7 composite score (maximum of 102.32 points). mNIS+7 composite total score range= -22.32 to 346.32. Higher score indicated a lower function. LS mean and SE were analyzed using MMRM. As pre-specified in the protocol, the efficacy of eplontersen was to be assessed by comparing participants enrolled in the eplontersen arm only with the external placebo group. There was no statistical comparison planned between the inotersen arm and the eplontersen-treated/external placebo group arms.
Time Frame: Baseline, Week 35
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Eplontersen | External Placebo
Number analyzed (Participants) | 138 | 55
scores on a scale | 0.6795 (1.9073) | 10.0337 (1.8544)
Statistical Analysis 1: Comparison: Eplontersen vs External Placebo; Test type: Superiority; p = 0.00012203, MMRM; Difference in LS Mean = -9.3542, 95% CI 2-sided [-13.8691 to -4.8394]

6. Secondary Outcome: Change From Baseline in Norfolk QOL-DN at Week 35
Description: as for outcome 2
Time Frame: Baseline, Week 35
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Groups:
- Placebo External Control: Participants in the external placebo arm received 3 SC doses of placebo during Week 1, followed by once-weekly SC administration for 64 weeks of the NEURO-TTR study.
Arm/Group | Eplontersen | Placebo External Control
Number analyzed (Participants) | 130 | 57
scores on a scale | -3.6306 (2.0678) | 8.1896 (2.0730)
Statistical Analysis 1: Comparison: Eplontersen vs Placebo External Control; Test type: Superiority; p = 0.00001873, MMRM; Difference in LS Mean = -11.8202, 95% CI 2-sided [-16.8927 to -6.7477]

7. Secondary Outcome: Change From Baseline in Neuropathy Symptom and Change (NSC) Score at Weeks 35 and 66
Description: NSC score is a questionnaire composed of 38 questions divided into 5 domains: muscle weakness, sensory (hypo/loss of sensation), sensory (paresthesia, hyper sensation), autonomic (gastrointestinal & urinary incontinence), & autonomic (non-GI/non-urinary incontinence)]. Answers to questionnaire are yes/no and if yes, then degree of severity is graded as 1 (slight +), 2 (moderate ++) and 3 (severe +++). 0=no symptom. NSC total score is a sum of scores across all 5 domains. Total score= 0-114. Higher scores=more neuropathy symptoms. LS mean and SE were analyzed using MMRM. As pre-specified in the protocol, the efficacy of eplontersen was to be assessed by comparing participants enrolled in the eplontersen arm only with the external placebo group. There was no statistical comparison planned between the inotersen arm and the eplontersen-treated/external placebo group arms.
Time Frame: Baseline, Week 35, Week 66
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Eplontersen | Placebo External Control
Number analyzed (Participants) | 141 | 57
scores on a scale
  At Week 35 | 0.79 (0.867) | 4.73 (0.870)
  At Week 66 | -0.03 (0.955) | 8.18 (0.962)
Statistical Analysis 1: Comparison: Eplontersen vs Placebo External Control; Week 35; Test type: Superiority; p = 0.00052447, MMRM; Difference in LS Mean = -3.94, 95% CI 2-sided [-6.08 to -1.80]
Statistical Analysis 2: Comparison: Eplontersen vs Placebo External Control; Week 66; Test type: Superiority; p = 0.00000001, MMRM; Difference in LS Mean = -8.21, 95% CI 2-sided [-10.65 to -5.76]

8. Secondary Outcome: Change From Baseline in the Physical Component Summary (PCS) Score of the 36-Item Short Form Survey (SF-36) at Week 65
Description: SF-36 comprises 36 items that yield 8 subscales and 2 summary measures (PCS and Mental component summary [MCS]). Multi-item subscales (35 items) includes: physical function=10 items, role physical =4 items, bodily pain=2 items, general health=5 items, vitality=4 items, social functioning=2 items, role emotional =3 items and mental health=5 items. 8 subscales are scored from 0-100. Higher scores indicate better health. 8 subscales are aggregated into a PCS score ranging from 0-100. Higher scores indicate better health. LS mean and SE were analyzed using MMRM. As pre-specified in the protocol, the efficacy of eplontersen was to be assessed by comparing participants enrolled in the eplontersen arm only with the external placebo group. There was no statistical comparison planned between the inotersen arm and the eplontersen-treated/external placebo group arms.
Time Frame: Baseline, Week 65
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Eplontersen | Placebo External Control
Number analyzed (Participants) | 136 | 50
scores on a scale | 0.851 (0.7913) | -4.455 (0.8338)
Statistical Analysis 1: Comparison: Eplontersen vs Placebo External Control; Test type: Superiority; p = 0.00000558, MMRM; Difference in LS Mean = 5.305, 95% CI 2-sided [3.195 to 7.416]

9. Secondary Outcome: Change From Baseline in Polyneuropathy Disability (PND) Score at Week 65
Description: PND is a 5-stage scoring system. PND score is defined as I=sensory disturbances in limbs without motor impairment; II=difficulty walking without the need of a walking aid; IIIa=one stick or one crutch required for walking; IIIb=two sticks or two crutches needed; IV=wheelchair required or patient confined to bed. For analysis, no impairment is scored as 0, I is scored as 1, II as 2, IIIa as 3, IIIb as 4 and IV as 5. Lower scores indicate greater ambulatory function. LS mean and SE were analyzed using MMRM. As pre-specified in the protocol, the efficacy of eplontersen was to be assessed by comparing participants enrolled in the eplontersen arm only with the external placebo group. There was no statistical comparison planned between the inotersen arm and the eplontersen-treated/external placebo group arms.
Time Frame: Baseline, Week 65
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Eplontersen | Placebo External Control
Number analyzed (Participants) | 134 | 51
scores on a scale | 0.1 (0.07) | 0.3 (0.07)
Statistical Analysis 1: Comparison: Eplontersen vs Placebo External Control; Test type: Superiority; p = 0.02407897, MMRM; Difference in LS Mean = -0.2, 95% CI 2-sided [-0.4 to -0.0]

10. Secondary Outcome: Change From Baseline in Modified Body Mass Index (mBMI) at Week 65
Description: mBMI is defined as body mass index in kilograms per square meter (kg/m^2) multiplied by serum albumin in grams per liter (g/L). As pre-specified in the protocol, the efficacy of eplontersen was to be assessed by comparing participants enrolled in the eplontersen arm only with the external placebo group. There was no statistical comparison planned between the inotersen arm and the eplontersen-treated/external placebo group arms.
Time Frame: Baseline, Week 65
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kilogram(kg)/metre(m)^2*gram(g)/litre(L)
Arm/Group | Eplontersen | Placebo External Control
Number analyzed (Participants) | 130 | 49
kilogram(kg)/metre(m)^2*gram(g)/litre(L) | -8.0655 (10.3786) | -90.7645 (10.9465)
Statistical Analysis 1: Comparison: Eplontersen vs Placebo External Control; Test type: Superiority; p = 0.00000020, MMRM; Difference in LS Mean = 82.6991, 95% CI 2-sided [54.6431 to 110.7551]

ADVERSE EVENTS:
Time Frame: Week 1 to Week 85
Description: Safety Set (SS) included all participants who were randomized and received at least 1 injection of eplontersen or inotersen.
Groups:
- Inotersen (Prior to Switch): Participants received inotersen, 300 mg, SC, once weekly from Week 1 through Week 34.
- Inotersen to ION-682884 (After Switch): Participants received eplontersen, 45 mg, SC, once every 4 weeks from Week 37 to Week 81.
Arm/Group | Eplontersen | Inotersen (Prior to Switch) | Inotersen to ION-682884 (After Switch)
All-Cause Mortality (participants affected / at risk) | 4/144 | 0/24 | 0/20
Serious Adverse Events (participants affected / at risk) | 27/144 | 3/24 | 3/20
Other Adverse Events (participants affected / at risk) | 131/144 | 24/24 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eplontersen (N=144) | Inotersen (Prior to Switch) (N=24) | Inotersen to ION-682884 (After Switch) (N=20)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Bradyarrhythmia (Cardiac disorders) | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Osteomyelitis chronic (Infections and infestations) | 0 | 1 | 0
Burns third degree (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Clostridium test positive (Injury, poisoning and procedural complications) | 1 | 0 | 0
Glomerular filtration rate decreased (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Syncope (Nervous system disorders) | 3 | 0 | 0
Cerebral haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Metabolic encephalopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Nephroangiosclerosis (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eplontersen (N=144) | Inotersen (Prior to Switch) (N=24) | Inotersen to ION-682884 (After Switch) (N=20)
Anaemia (Blood and lymphatic system disorders) | 7 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 4 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 8 | 2 | 0
Cataract (Eye disorders) | 8 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 28 | 1 | 1
Nausea (Gastrointestinal disorders) | 14 | 5 | 0
Vomiting (Gastrointestinal disorders) | 11 | 4 | 1
Oedema peripheral (General disorders) | 13 | 0 | 2
Fatigue (General disorders) | 8 | 6 | 2
Injection site pain (General disorders) | 5 | 3 | 0
Injection site erythema (General disorders) | 5 | 8 | 0
Pyrexia (General disorders) | 4 | 7 | 0
Injection site bruising (General disorders) | 2 | 5 | 0
Peripheral swelling (General disorders) | 2 | 0 | 1
Chills (General disorders) | 1 | 5 | 0
Pain (General disorders) | 1 | 2 | 0
Injection site swelling (General disorders) | 0 | 3 | 0
Immunisation reaction (Immune system disorders) | 13 | 1 | 0
Urinary tract infection (Infections and infestations) | 26 | 2 | 4
COVID-19 (Infections and infestations) | 47 | 1 | 5
Nasopharyngitis (Infections and infestations) | 9 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 9 | 1 | 0
Influenza (Infections and infestations) | 7 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 10 | 2 | 2
Thermal burn (Injury, poisoning and procedural complications) | 6 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 2 | 0
Alanine aminotransferase increased (Investigations) | 5 | 2 | 0
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 9 | 0 | 1
Weight decreased (Investigations) | 4 | 0 | 1
Glomerular filtration rate Decreased (Investigations) | 3 | 4 | 2
Platelet count decreased (Investigations) | 2 | 2 | 0
Vitamin A deficiency (Metabolism and nutrition disorders) | 17 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 5 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 5 | 0
Dizziness (Nervous system disorders) | 11 | 0 | 1
Headache (Nervous system disorders) | 9 | 5 | 1
Neuralgia (Nervous system disorders) | 5 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 6 | 1 | 1
Depression (Psychiatric disorders) | 5 | 0 | 2
Anxiety (Psychiatric disorders) | 4 | 0 | 2
Proteinuria (Renal and urinary disorders) | 12 | 1 | 1
Urinary retention (Renal and urinary disorders) | 6 | 0 | 1
Albuminuria (Renal and urinary disorders) | 2 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 7 | 2 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 6 | 2 | 0
Hypotension (Vascular disorders) | 5 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/84/NCT04136184/Prot_SAP_000.pdf